CLINICAL TRIAL: NCT07176598
Title: Case Report: Misdiagnosed Primary Intramuscular Hydatid Cyst of the Deltoid Muscle in a Male Patient
Brief Title: Rare Case of Misdiagnosed Primary Intramuscular Hydatid Cyst of the Deltoid Muscle
Acronym: RPHC-Deltoid
Status: Completed | Type: Observational
Sponsor: Al-Shahba Specialized Hospital (Other)
Responsible Party: Principal Investigator, Mohanad Nasani, Dr. Mohanad Nasani, Al-Shahba Specialized Hospital
Other Study IDs: RC-Hydatid-2025-001
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Primary Intramuscular Hydatid Cyst Hydatid Disease (Echinococcosis)
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This case report describes a rare parasitic cyst called a hydatid cyst located in the shoulder muscle (deltoid) of a 29-year-old male. The patient initially presented with a painless, gradually enlarging swelling over the left shoulder. It was misdiagnosed as a synovial cyst and treated with corticosteroids, which caused local inflammation and purulent discharge. Blood tests for Echinococcus antibodies were negative. Ultrasound and MRI revealed a well-defined intramuscular cyst confined to the deltoid muscle. Surgical excision confirmed the diagnosis, and the patient received postoperative albendazole therapy for three months. Follow-up showed complete healing, restoration of shoulder function, and no recurrence. This case highlights the importance of considering hydatid disease in unusual muscle locations, particularly in endemic areas, to avoid misdiagnosis and ensure proper treatment.

DETAILED DESCRIPTION:
This report presents a rare case of a primary intramuscular hydatid cyst confined to the deltoid muscle in a 29-year-old male. The patient had a seven-month history of a gradually enlarging swelling in the left shoulder. Initially misdiagnosed as a synovial cyst, he received corticosteroid injection, which led to pain, erythema, and purulent discharge. Physical examination revealed a 10 cm fluctuant mass over the posterolateral deltoid. Serology for Echinococcus antibodies was negative. Ultrasound showed a well-defined, anechoic intramuscular cyst measuring 7 × 8 × 10 cm. MRI confirmed a fluid-filled cyst confined to the deltoid muscle, without involvement of bone, tendon, or joint structures. Under local anesthesia, the cyst was completely excised, and the cavity was irrigated with 10% povidone-iodine. Histopathology confirmed a non-fertile hydatid cyst (Echinococcus granulosus) without malignancy. Postoperative therapy included albendazole 400 mg daily for three months. Follow-up at six weeks showed complete wound healing, full shoulder function, and no recurrence. This case underscores the diagnostic challenges of intramuscular hydatid cysts, especially with negative serology, and highlights the importance of imaging, histopathology, and careful surgical management in endemic regions.

ELIGIBILITY:
Inclusion Criteria:

Male patient Age 18 years or older Diagnosed with primary intramuscular hydatid cyst of the deltoid muscle

Exclusion Criteria:

Patients with cysts in other organs (liver, lungs) Patients with systemic infection or immunocompromised status Patients who did not undergo surgical excision

-

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A single 29-year-old male patient diagnosed with primary intramuscular hydatid cyst of the deltoid muscle. The patient underwent surgical excision and postoperative albendazole therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Complete recovery of shoulder function without recurrence | 6 weeks postoperatively
  Monitoring for surgical site infection, serological status, and general patient well-being following treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Shahbaa Specialized Hospital, Aleppo, Syria